CLINICAL TRIAL: NCT04077099
Title: A Phase 1/2 Study of REGN5093 in Patients With MET-Altered Advanced Non-Small Cell Lung Cancer
Brief Title: A Study of REGN5093 in Adult Patients With Mesenchymal Epithelial Transition Factor (MET)-Altered Advanced Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R5093-ONC-1863; 2019-001908-38 (EudraCT Number); 2023-506248-18-00 (EU CTIS Number)
Record Dates: First submitted 2019-08-13; First posted 2019-09-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: NSCLC
Keywords: MET (mesenchymal-epithelial transition factor); HGF (Hepatocyte Growth Factor); NSCLC (non-small cell lung cancer); MET-altered advanced; Unresectable; Metastatic disease
MeSH Terms: conditions — Deafness, Autosomal Recessive 39; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- REGN5093 (Experimental): Monotherapy in dose escalation cohorts (phase 1) followed by an expansion phase (phase 2)
  Interventions: Drug: REGN5093

INTERVENTIONS:
Drug: REGN5093 — Intravenous (IV) infusion. There will be a series of dose escalation cohorts followed by an expansion phase.

SUMMARY:
This study will evaluate REGN5093 for the treatment of Non-Small Cell Lung Cancer (NSCLC) with MET alteration. The main purpose of this study is to determine the safety, tolerability, and effectiveness of REGN5093.

The study has two phases. The main goal of Phase 1 is to determine a safe dose(s) of REGN5093. The main goal of phase 2 of the study is to use the REGN5093 drug dose(s) found in Phase 1 to see how well REGN5093 works to shrink tumors.

The study is looking at several other research questions, including:

* Side effects that may be experienced by people taking REGN5093
* How REGN5093 works in the body
* How much REGN5093 is present in the blood
* To see if REGN5093 works to reduce or delay the progression of cancer
* How long it takes REGN5093 to work in the body

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed advanced NSCLC that is unresectable or metastatic as described in the protocol
2. Willing to provide tumor tissue as described in the protocol
3. Documented presence of MET alteration as described in the protocol.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Adequate organ and bone marrow function as described in the protocol

Key Exclusion Criteria:

1. Has received treatment with an approved systemic therapy or has participated in any study of an investigational agent or investigational device within 2 weeks as described in the protocol
2. Has not yet recovered from any acute toxicities resulting from prior therapy with certain exceptions as described in the protocol
3. Has received radiation therapy or major surgery within 14 days as described in the protocol
4. Untreated or active primary brain tumor, central nervous system (CNS) metastases, leptomeningeal disease or spinal cord compression as defined in the protocol
5. Uncontrolled infection as described in the protocol

Note: Other protocol defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2032-04-22 (Estimated); Study Completion 2032-04-22 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Dose Limiting Toxicities (DLTs) | Up to 21 days
  Phase 1/Dose escalation
Incidence and severity of treatment-emergent adverse events (TEAEs) | Through study completion, an average of 12 years
  Phase 1/Dose escalation
Incidence and severity of adverse events of special interest (AESIs) | Through study completion, an average of 12 years
  Phase 1/Dose escalation
Incidence and severity of serious adverse events (SAEs) | Through study completion, an average of 12 years
  Phase 1/Dose escalation
Incidence and severity of grade ≥3 laboratory abnormalities | Through study completion, an average of 12 years
  Phase 1/Dose escalation
REGN5093 concentrations in serum over time | Through study completion, an average of 12 years
  Phase 1/Dose escalation
Objective response rate (ORR) per RECIST 1.1 | Through study completion, an average of 12 years
  Phase 2/Dose expansion

SECONDARY OUTCOMES:
ORR per RECIST 1.1 | Through study completion, an average of 12 years
  Phase 1/Dose escalation
Incidence and severity of TEAEs | Through study completion, an average of 12 years
  Phase 2/Dose expansion
Incidence and severity of AESIs | Through study completion, an average of 12 years
  Phase 2/Dose expansion
Incidence and severity of SAEs | Through study completion, an average of 12 years
  Phase 2/Dose expansion
Incidence and severity of grade ≥3 laboratory abnormalities | Through study completion, an average of 12 years
  Phase 2/Dose expansion
REGN5093 Pharmacokinetics (PK) | Through study completion, an average of 12 years
  Phase 2/Dose expansion
REGN5093 concentrations in serum over time | Through study completion, an average of 12 years
  Phase 2/Dose expansion
Duration of response (DOR) per RECIST 1.1. | Through study completion, an average of 12 years
  Phase 1 and 2
Disease control rate (DCR) per RECIST 1.1. | Through study completion, an average of 12 years
  Phase 1 and 2
Progression free survival (PFS) per RECIST 1.1. | Through study completion, an average of 12 years
  Phase 1 and 2
Overall survival (OS) | Through study completion, an average of 12 years
  Phase 1 and 2
Time to response (TTR) per RECIST 1.1 | Through study completion, an average of 12 years
  Phase 1 and 2
Incidence of anti-drug antibodies (ADA) to REGN5093 | Through study completion, an average of 12 years
  Phase 1 and 2
Titer of ADA to REGN5093 | Through study completion, an average of 12 years
  Phase 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (33):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Irvine Medical Center - Bldg 56, RT81, Rm 241, Orange, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Moffitt Cancer Center - McKinley Drive, Tampa, Florida
  - University of Kentucky, Markey Cancer Center Clinical Research Organization, Lexington, Kentucky
  - DNU_Massachusetts General Hospital_DNU, Boston, Massachusetts
  - Dana Farber Harvard Cancer Center Consortium, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Cancer Institute, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh UPMC - Clinical Research Services, Pittsburgh, Pennsylvania
  - Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- France (6):
  - Centre Georges Francois Leclerc, Dijon, Bourgogne-Franche-Comté
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes, Bretange
  - Centre Francois Baclesse (CFB), Caen, Normandy
  - Institut Bergonie, Bordeaux, Nouvelle-Aquitaine
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Centre Hospitalier Regional Universitaire (CHRU) Montpellier Arnaud de Villeneuve, Montpellier
- South Korea (9):
  - National Cancer Center, Gyeonggi-do, Gyeonggi-do
  - The Catholic University Of Korea St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Haeundae Paik Hospital, Pusan, Gyeongsangnam-do
  - Pusan National University Hospital, Busan
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seol St. Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * has the legal authority to share the data, and
  * has ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/